CLINICAL TRIAL: NCT05727384
Title: Reducing Inflammation for Greater Health Trial: The RIGHT Study
Brief Title: Improving Physical Function in Older Adults Using an Anti-inflammation Drug: The RIGHT Study
Acronym: RIGHT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anne B. Newman (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor-Investigator, Anne B. Newman, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19030225
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Inflammation; Frailty
MeSH Terms: conditions — Inflammation; Frailty | interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clazakizumab (Experimental): Participants received Clazakizumab 5 mg as a subcutaneous injection every 4 weeks for 24 weeks
  Interventions: Drug: Clazakizumab
- Placebo (Placebo Comparator): Participants received Clazakizumab placebo as a 5 mg subcutaneous injection every 4 weeks for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clazakizumab — 5 mg, subcutaneous injection, every 4 weeks for 24 weeks
  Arms: Clazakizumab
Drug: Placebo — 5 mg, subcutaneous injection, every 4 weeks for 24 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the effects of inflammation-lowering therapy on mobility and disability in older adults. The main questions it aims to answer are:

* Will therapy improve walking speed/pace?
* Will therapy improve levels of blood inflammation markers and other indicators of physical, cognitive and immune function?

Participants will be asked to receive injections of drug or placebo every 4 weeks for 24 weeks. They will also be asked to undergo testing that assesses physical function, thinking ability and brain health, breathing capacity, and blood vessel stiffness, and will have blood samples collected to measure immune function and to create a bank of samples for future testing. Comparisons will be made between those who receive drug and those who receive placebo.

DETAILED DESCRIPTION:
The primary objective of this trial is to assess the impact of inflammation-lowering therapy with clazakizumab 5 mg/month on speed when walking 400 meters in older adults. The investigators hypothesize that participants treated with clazakizumab will see a larger 6-month improvement in their pace on a 400-meter walk than those provided placebo.

The aims of the study will be to:

* To test the effect of clazakizumab 5 mg/month for 6 months on walking speed during a 400- meter corridor walk in adults 70 years of age and older with baseline levels of IL-6 ≥ 2.0 pg/ml and < 30 pg/ml
* To assess the effect of clazakizumab 5 mg/month on serum levels of free interleukin (IL-6), circulating C-reactive protein (CRP), and other inflammatory markers
* To assess the effect of clazakizumab 5 mg/month on oxygen utilization (VO2) during submaximal steady-state walking in adults 70 years of age and older with baseline levels of IL-6 ≥ 2.0 pg/ml and < 30 pg/ml, physical function, physical activity, perceived fatigability (overall, by questionnaire and in association with preferred and fixed speed walking), cognition, body weight, blood pressure, vascular stiffness, endothelial function, kidney function and immune function
* To determine the safety and tolerability of clazakizumab 5 mg/month

This study will randomize 60 community living men and women 70 years of age and older who have mildly elevated IL-6 at baseline (≥ 2.0 pg/ml and < 30.0 pg/ml). Interested individuals will undergo telephone and in-person screening visits (two) to determine eligibility (blood will be collected to measure IL-6, height and weight will be measured, a 4m walk test will be administered to determine gait speed, and a review of medical history, medications, a physical exam, and blood safety labs will be conducted to ensure safety to proceed/eligibility). Randomization to study drug or placebo will take place within 60 days of the first in-person screening visit and subsequent injections will take place every 4 weeks for 24 weeks. Participants will undergo physical function testing (400m walk, preferred & fixed speed walk on a treadmill with oxygen consumption measurement, short physical performance battery, grip strength, actigraphy), cognitive testing, and aortic pulse wave velocity and endothelial function testing. Height, weight and pulse will be measured. Participants will complete questionnaires to assess demographics, physical activity level, fatigability, sleep quality, pain and depression. Blood will be collected/processed to measure immune function and stored frozen to create a biorepository of samples (serum, plasma, buffy coat) for future testing. Participants will be monitored for safety in between injection visits and for 5 months following the final in-person research visit.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged ≥ 70 years at time of randomization
* Gait speed ≥ 0.44 m/sec to < 1.0 m/sec or BMI ≥ 28 kg/m2
* IL-6 level ≥ 2.0 pg/ml but < 30.0 pg/ml
* Self-reported difficulty walking ¼ mile or climbing 10 steps
* Self-reported ability to walk 400 meters (about 2-3 blocks), unassisted
* Self-reported vaccinations for COVID-19, Influenza and pneumococcal pneumonia up to date per current CDC guidelines

Exclusion Criteria:

* Advanced neurologic disorder such as dementia, Parkinson's disease, amytrophic lateral sclerosis, or multiple sclerosis that would impact the ability to improve on functional assessments
* Resident in a nursing home
* Severe hearing or vision loss that would impair participant's ability to complete questionnaires or follow oral instructions, and which may limit feasibility of performing functional assessments
* Acute infections (including but not limited to common cold virus, shingles virus, bronchitis, skin infection, urinary tract infection, tooth abscess) within 60 days of randomization
* Chronic infection (including but not limited to):

  * History of active TB or evidence of latent TB based on a positive PPD skin test, positive Quantiferon TB-Gold test, or a history of old or latent TB on chest x-ray
  * History of Hepatitis B or Hepatitis C
  * Previous diagnosis of Human Immunodeficiency Virus (HIV) or Acquired ImmunoDeficiency Syndrome (AIDS)
* Inflammatory or autoimmune disease (including but not limited to rheumatoid arthritis, lupus, or inflammatory bowel disease, such as ulcerative colitis or Crohn's disease)
* Immunization with a live/attenuated vaccine within 2 months prior to randomization (e.g., viral: measles vaccine, mumps vaccine, rubella vaccine, live attenuated influenza vaccine, live attenuated chicken pox or shingles vaccine, smallpox vaccine, oral polio vaccine (Sabin), rotavirus vaccine, and yellow fever vaccine. Bacterial: BCG vaccine, oral typhoid vaccine and epidemic typhus vaccine)
* Current use of chronic immune modulating medications such as corticosteroids, monoclonal antibodies, janus kinase inhibitors, calcineurin inhibitors, mTOR inhibitors, IMDH inhibitors, or biologics
* Admitted for an overnight hospitalization in the last 6 months
* Open-chest heart surgery (including, but not limited to, coronary artery bypass graft surgery or aortic valve surgery) in the past 6 months
* Anticipating major surgery (including, but not limited to, chest, abdomen, or joint surgery) in the next 6 months
* Deep vein thrombosis or pulmonary embolus in the past 6 months
* Severe lung disease or heart disease that requires oxygen use anytime during the day (including, but not limited to, use only during activity, use only at night or use all day)
* Tobacco use (including cigarettes, cigar, pipe, or vaping) or inhaled cannabis in the past 6 months
* Current consumption of > 14 alcoholic drinks per week
* History of substance abuse including cocaine, methamphetamine, opioids, or narcotics; any use of cannabis
* Uncontrolled diabetes, noncompliant with treatment or fasting glucose > 250 mg/dL
* Cancer: Stage 1 cancer (including melanoma skin cancers) within the past 5 years, other than adequately treated (fully excised and recovered from surgery based on the judgement of a study MD) basal and/or squamous cell skin cancer, or stage 2 or stage 3 cancer within 10 years, or any history of stage 4 (metastatic) cancer
* Inability to get a normal systolic blood pressure reading (between 100-180) at two consecutive visits prior to randomization (must be at least 1 day apart)
* ALT, AST, or Total Bilirubin > Upper Limit of Normal (ULN)
* Absolute Neutrophil Count outside normal range or < 1.5 x109/L
* White Blood Count outside normal range
* Platelet count outside normal range or < 125 x109/L
* Hemoglobin <10 g/dL
* Total Cholesterol > 300 mg/dL or Triglycerides > 400 mg/dL
* Dialysis treatment or chronic renal insufficiency defined as CKD-EPI eGFR < 25 ml/min/(1.73) m2
* History of diverticular disease or GI perforation
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Current use of Warfarin (Coumadin, Jantoven)
* Unable or unwilling to provide informed consent
* Current participation in another interventional study (including trials of exercise, diet, or investigational drugs)
* A psychiatric disorder that is impairing ability to consent or comply with requirements of the trial
* Residence or travel outside of the study area for more than one month during the study or planning to move out of the area in the next six months.
* Other conditions which at the discretion of a study physician investigator which would make participation unsafe or inappropriate (logistic, behavioral, medical)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Speed of Walking 400 Meters from Baseline to 24 Weeks | From enrollment (randomization/first drug injection visit) to the final research assessment visit (4 weeks after final drug injection visit or 24 weeks after enrollment)
  Assess effect of Clazakizumab versus placebo on speed of walking 400 meters (meters/second) from baseline to 24 weeks

SECONDARY OUTCOMES:
Mean Change in Oxygen Consumption While Walking from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess effect of Clazakizumab versus placebo on change of oxygen consumption (VO2 measured as ml/kg/min) with fixed speed walking on treadmill from baseline to 24 weeks
Mean Change in Physical Function using the Short Physical Performance Battery (SPPB) Score from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess effect of Clazakizumab versus placebo on change in Short Physical Performance Battery score (0-12 scale, higher score better) from baseline to 24 weeks
Mean Change in Muscle (Grip) Strength from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in muscle grip strength (kg) from baseline to 24 weeks
Mean Change in Fatigue Level using the Pittsburgh Fatigability Score (PFS) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in Pittsburgh Fatigability Score (0-100 scale, higher score indicates greater mental & physical fatigue) from baseline to 24 weeks
Mean Change in Vascular Stiffness using Aortic Pulse Wave Velocity (APWV) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in Aortic Pulse Wave Velocity (cm/sec) from baseline to 24 weeks
Mean Change in Peripheral Microvascular Endothelial Function using Peripheral Arterial Tonometry (EndoPat) from baseline to 24 weeks. | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in EndoPat derived indices: 1) reactive hyperemia index (RHI is a ratio; higher values indicate greater vessel vasodilator capacity) and 2) augmentation index (AI%; lower values indicate greater vessel elasticity) from baseline to 24 weeks.
Mean Change in Cognitive Function using the Montreal Cognitive Assessment (MoCA) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the Montreal Cognitive Assessment score (0-30 scale, higher is better) from baseline to 24 weeks
Mean Change in Cognitive Function using the California Verbal Learning Test (CVLT) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the number correct for short word recall and long word recall (0-16 words recalled, each of 5 trials, higher is better), and the number of word intrusions/repetitions using the California Verbal Learning Test from baseline to 24 weeks
Mean Change in Cognitive Function using the Digit Symbol Substitution Test (DSST) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the number correct in 90 seconds (higher is better) on the Digit Symbol Substitution Test from baseline to 24 weeks
Mean Change in Cognitive Function using the Trails Making B (Trails B) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the time to complete (seconds, lower is better) Trails Making Test B from baseline to 24 weeks
Mean Change in Inflammatory Biomarker Interleukin 6 (IL-6) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on Interleukin 6 (pg/mL) from Baseline to 24 weeks
Mean Change in Inflammatory Biomarker C-Reactive Protein (CRP) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on C-Reactive Protein (mg/dL) from Baseline to 24 weeks
Assess Safety and Tolerability of Clazakizumab by Monitoring Adverse Events (AEs) and Serious Adverse Events (SAEs) From Baseline to 44 Weeks | AEs and SAEs assessed weekly after randomization/first drug injection visit, one week after drug visits 2-6, at the final research assessment visit (24 weeks after baseline), and every 4 weeks for 20 weeks after the final research assessment visit
  Assess the number of study participants reporting Adverse Events and Severe Adverse Events following the drug injection visits, at the final research assessment visit (24 weeks after baseline), and every 4 weeks for 20 weeks after the final research assessment visit
Assess Safety and Tolerability of Clazakizumab by Monitoring Safety Laboratory Values From Baseline to 24 Weeks | assessed weekly after randomization/first drug injection visit, one week after drug visits 2-6, at the final research assessment visit (24 weeks after baseline)
  Compare the percent of participants (Clazakizumab versus placebo) with safety laboratory values for total white blood cell count, absolute neutrophil count, platelet count, liver function (alanine aminotransferase, aspartate aminotransferase and bilirubin, and lipids (total, HDL, and LDL cholesterol and triglycerides) outside of the normal range (as specified in the study protocol) to safely administer the study drug following the drug injection visits, and at the final research assessment visit (24 weeks after baseline).
Assess Tolerability of Clazakizumab by Monitoring Adherence to Drug Administration From Baseline to 20 Weeks | Assessed at the time of the drug injection visits from baseline (randomization/first injection) through drug visits 2-6.
  Tolerability will be assessed as adherence to the protocol expressed as a percentage of doses received and percentage of drug dosing visits attended in those receiving Clazakizumab versus placebo assessed following each drug injection visit (randomization/first drug injection visit and drug visits 2-6) line).
Change in Dementia Biomarker Levels from Baseline to 24 Weeks. | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on dementia biomarker levels as measured in peripheral blood, from baseline to 24 weeks. These include 1) Aβ42 and Aβ40 amyloid, 2) phosphorylated tau protein neurofilament light chain, and 3) glial fibrillary acidic protein (all in pg/ml).

OTHER OUTCOMES:
Mean Change in Physical Activity Level using the Community Health Activities Model Program for Seniors (CHAMPS) Questionnaire from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change estimated kilocalories/kg/week and hours of moderate activity per week assessed by the Community Health Activities Model Program for Seniors from baseline to 24 weeks
Mean Change in Physical Activity Level as Assessed by Actigraphy from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess effect of Clazakizumab versus placebo on change in mean time engaged in moderate to vigorous physical activity (MVPA) in minutes/week measured with actigraphy from baseline to 24 weeks
Mean Change in Quality of Life using the Short Form 36 (SF-36) Health Survey from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the Short Form-36 Health Survey score (0-100 scale, higher is better) from baseline to 24 weeks
Mean Change in Depression/Depressive Symptomatology using the Center for Epidemiologic Studies Depression Scale (CES-D) Short Form from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change Center for Epidemiologic Studies Depression Scale score (0-60 scale, higher is worse) from baseline to 24 weeks
Mean Change in Sleep-Related Impairment using the Patient-Reported Outcomes Measurement Information System (PROMIS) from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in Patient-Reported Outcomes Measurement Information System sleep-related impairment (8-40 scale, higher is worse) from baseline to 24 weeks
Mean Change in Disability using the Physical Subscale of Short Form 36 (SF-36) Health Survey from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in disability using the physical subscale of the Short Form 36 Health Survey score (0-100 scale, higher is better) from baseline to 24 weeks
Change in Frequency of Immune B Cell, T Cell and Memory B Cell Subsets from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the frequency (percent) of immune cell subsets (T cells, B cells, Memory B cells) using flow cytometry from Baseline to 24 weeks
Change in Counts of Immune B Cell, T Cell and Memory B Cell Subsets from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in the counts (cells/microliter) of B cell, T cell and memory B cell subsets measured by flow cytometry from Baseline to 24 weeks
Change in CD-8 T Cell Function from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on change in CD-8 T cell function in response to ex vivo stimulation measured by flow cytometry from Baseline to 24 weeks
Mean Change in Inflammatory Cytokines using a 36-Plex Kit from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on 36 cytokines (pg/mL) included in the Myriad V-PLEX Plus Human Cytokine 36-Plex kit from Baseline to 24 weeks
Assess the effect of Clazakizumab versus placebo on brain structure, including white matter lesions, from baseline to 24 weeks. | Baseline (randomization/first drug injection visit) to teh final research assessment visit (24 weeks after baseline)
  Brain structure will be assessed with a high-resolution, 3-dimensional MPRAGE structural MRI scan (~6 min). Values and units: Voxels (mm3). Change in voxels for whole brain and hippocampus before and after treatment
  White matter hyperintensities will be assessed with a T2 3d FLAIR scan (~7 minutes). Values and units: Voxels (mm3) and change in voxels.
Change in Brain Function from Baseline to 24 Weeks. | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline)
  Assess the effect of Clazakizumab versus placebo on brain function from baseline to 24 weeks with echoplanar MRI imaging of blood oxygen level-dependent (BOLD) response while resting (~10 min).
  Values and units: Pearson's correlation coefficient. Change in correlation before and after treatment.
Change in Brain Connectivity from Baseline to 24 weeks. | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline).
  Assess the effect of Clazakizumab versus placebo on structural connectivity from baseline to 24 weeks with a diffusion weighted MRI scan (~12min).
  Values and units:
  1. Number of tracts
  2. Length of tracts (mm)
  3. Fractional Anisotropy (FA): A measure of the degree to which water diffusion is directional within a voxel, reflecting the alignment of white matter fibers. Higher FA indicates more organized white matter. No units. Change in FA values will be assessed before and after treatment.
Change in Brain Blood Flow from Baseline to 24 Weeks | From baseline (randomization/first drug injection visit) to the final research assessment visit (24 weeks after baseline).
  Assess the effect of Clazakizumab versus placebo from baseline to 24 weeks on brain connectivity via blood flow as assessed with brain MRI arterial spin labeling (ASL) (~6 min).
  Values and units: mL/100 g/min before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne B. Newman, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Health Studies Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data to be shared include clinical characteristics pre-and post-intervention, a data dictionary, and documentation of analytical tools used in data processing (e.g., normalization, unit conversion, etc.).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available approximately 6 months after the study describing the data is accepted for publication (seminal publication). The data will be made available for an indefinite period of time to be determined by the study Principal Investigator.
Access Criteria: All individuals will be required to enter into a Data Use Agreement that a) acknowledges that the data will be stripped of identifying markers and unusual characteristics that might provide identification, (b) acknowledge that these data will only be used for research purposes, and (c) assure that the investigator will either destroy the raw data or return it to Dr. Newman (Study PI) when their research has been completed. Individuals will also be required to reference the seminal publication describing the data collection and acknowledge the source of funding.

REFERENCES:
- [Derived] Sattui SE, Bertolet M, Forman DE, Danielson ME, Yao S, Lopez OL, Glynn NW, Nadkarni NK, Sekikawa A, Bruno TC, Finkel T, Newman AB. The "Reducing Inflammation for Greater Health Trial (RIGHT)" Study-Concept, Rationale, and Design. J Am Geriatr Soc. 2026 Jan 10. doi: 10.1111/jgs.70272. Online ahead of print. PMID 41518612